CLINICAL TRIAL: NCT06626464
Title: A Phase 1 Clinical Study to Evaluate the Absorption, Metabolism and Excretion of [14C]MK-8189 in Healthy Adults
Brief Title: A Study of MK-8189 Human Absorption, Metabolism, and Excretion in Healthy Male Participants (MK-8189-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8189-010; MK-8189-010 (Other: MSD)
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carbon-14 radiolabeled [14C] MK-8189 (Experimental): Participants receive a dose of 4.5-mg immediate release (IR) (~ 50 μCi) orally on Day 1.
  Interventions: Drug: [14C]MK-8189

INTERVENTIONS:
Drug: [14C]MK-8189 — Oral administration

SUMMARY:
The purpose of this study is to learn what happens to MK-8189 in a healthy person's body over time.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria include but are not limited to the following:

* Is in good health based on medical history, physical examination, VS measurements, and ECGs performed before randomization.
* Has a BMI ≥19 and ≤32 kg/m2, inclusive, at screening

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Has a history of cancer.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from 0 to 24 hours (AUC0-24) of MK-8189 | Predose and postdose up to 24 hours
  Blood samples will be collected to determine the AUC0-24 of MK-8189.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the AUClast of MK-8189.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the AUC0-inf of MK-8189.
Maximum Concentration (Cmax) of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the Cmax of MK-8189.
Apparent Half Life (t½) of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the t1/2 of MK-8189.
Time to Reach Maximum Concentration (Tmax) of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the Tmax of MK-8189.
Amount Excreted (Ae) in Urine of MK-8189 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the Ae of MK-8189
%Dose Excreted in Urine of MK-8189 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the %dose of MK-8189
Amount Excreted (Ae) in Feces of MK-8189 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the Ae of MK-8189.
%Dose Excreted in Feces of MK-8189 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the %dose of MK-8189.
Metabolites in Plasma of MK-8189 | Predose and at designated timepoints up to Day 15
  Blood samples will be collected to determine the metabolites of MK-8189.
Metabolites in Urine of MK-8189 | Predose and at designated timepoints up to Day 15
  Urine samples will be collected to determine the metabolites of MK-8189.
Metabolites in Feces of MK-8189 | Predose and at designated timepoints up to Day 15
  Feces samples will be collected to determine the metabolites of MK-8189.

SECONDARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to ~ 28 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.
Number of Participants Discontinuing Study Treatment due to an AE | Up to ~ 28 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. For each arm, the number of participants experiencing an AE will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Labcorp Clinical Research Unit Inc. (Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com